CLINICAL TRIAL: NCT04005937
Title: Optimal Interstimulus Interval For Consecutive H-Reflex Responses In Patients With Spasticity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IstPMRTRH
Record Dates: First submitted 2019-06-30; First posted 2019-07-02 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Muscle Hypertonia; Reflex, Abnormal
Keywords: muscle spindle; H reflex; spasticity
MeSH Terms: conditions — Muscle Hypertonia; Reflex, Abnormal; Muscle Spasticity | interventions — H-Reflex

STUDY DESIGN:
Intervention Model Description: Effects of spasticity on consecutive H-reflex response in patients with hemiplegia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- H-reflex (Experimental): H-reflex with different interstimulus interval of the plegic side soleus muscle were tested
  Interventions: Diagnostic Test: H-reflex

INTERVENTIONS:
Diagnostic Test: H-reflex — Electrical stimulation of Group Ia afferent of muscle spindle

SUMMARY:
This study evaluates the optimal interstimulus interval for consecutive H-reflex responses in patients with spasticity.

DETAILED DESCRIPTION:
This study will include 15 patients with spastic stroke patients H-reflex with different interstimulus interval of the plegic side soleus muscle will be tested.

Subjects lay comfortably in the supine position on an examination bed. The subject will be asked not to contract the lower extremity muscles during the experiment. Surface EMG (SEMG) will be recorded from the plegic side soleus muscle using bipolar electrodes. These electrodes will be placed on the soleus muscle according to the SENIAM guideline.The reference electrode will be placed on medial malleolus. Prior to electrode placement, the skin will be shaved, lightly abraded, and cleaned with alcohol wipes. Self-adhesive, disposable, Ag-AgCl disc electrodes with a disc radius of 10 mm (KENDALL® Arbo; Coviden; Massachusetts, USA) will be used. To prevent the sway of electrode cables, it will be fixed to the body. SEMG and stimulator data will be obtained by using a data acquisition system (POWERLAB® ADInstruments Co, Oxford, United Kingdom). Sampling rate will be 10 kHz.

The recorded data will be processed and analyzed offline using LabChart7® Software Version V7.3.3 (PowerLab® system ADInstruments, Oxford, United Kingdom).

A cathode (5×5 mm) will be placed at the midpoint of popliteal fossa and an anode (10×10 cm) will be placed immediately proximal to the patella to evoke the H-reflex for monopolar stimulation of the posterior tibial nerve. A monophasic electrical current will be delivered as square pulses with a width of 1 ms by using a stimulator (FE155 Stimulator HC ADInstrument, Oxford UK). Taking into consideration study of Ozyurt et al, interstimulus interval will be selected as 10 seconds for determining the maximum H-reflex (Hmax). Then, Hmax and M-response (Mmax) will be determined.

We will be tested four different ISI (10s, 5s, 3s and 1s) for stroke patients in this study. The stimulus intensity for tested H-reflex will be selected as a constant stimulus strength that will be 50 percent of the Hmax.

Thirty consecutive stimuli will be delivered in separate sets for each tested ISI of 10, 5, 3 and 1s. The ISI sets will be tested in random order to negate any order effect. There will be a 15s of interval between sets.

SEMG recordings will be filtered using a bandpass filter from 5 to 500 Hz. Then the peak-to-peak (P-P) amplitudes of H-reflex will be measured then normalized using by two different methods to estimate H-reflex suppression due to consecutive stimuli. In the first method, P-P amplitude of the first H-reflex response will be used as a control, and P-P amplitude of the second H-reflex response will be normalized by using the control for each ISI set. Thus, HPP2 / HPP1 ratio will be calculated. Similar to the previous method, the first H-reflex response will be used as the control in the second method. Unlike the first method, not only the second H-reflex response, but the remaining 29 H-responses will be normalized to the first H-response. P-P amplitude of the 29 normalized H-reflex responses will be averaged and HPP29/HPP1 ratio will be calculated.

The peak-to-peak amplitude of the first H-reflex response will be measured then normalized to the Mmax (HPP1/Mmax) to compare H-reflexes between subjects and conditions.

ELIGIBILITY:
Inclusion Criteria:

* Cerebrovascular stroke
* Both sex

Exclusion Criteria:

* Duration after stroke is less than 20 days
* Lesions in calf skin
* Excessive spasticity (Ashworth 4) / Contracture (foot joint)
* Absent of soleus spasticity
* Peripheral nerve diseases / muscle diseases
* Absent of H-reflex
* Botulinum toxin injection within last 12 weeks
* Anxiety
* Patients with pain on test day

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-06-30 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
H-reflex suppression | 1 day
  Change in H-reflex amplitude throughout consecutive stimuli

CONTACTS AND LOCATIONS:
Overall Officials: Dilara Ekici, MD, Principal Investigator — stanbul Physical Medicine Rehabilitation Training and Research Hospital Istanbul
Locations (2):
- Turkey (Türkiye) (2):
  - stanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Bahçelievler
  - Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No